CLINICAL TRIAL: NCT05359861
Title: A Randomized Phase 2 Trial of Atezolizumab and Bevacizumab in Combination With SRF388 or Placebo in Patients With Untreated Locally Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: Trial of Atezolizumab and Bevacizumab With SRF388 or Placebo in Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRF388-201
Record Dates: First submitted 2022-04-14; First posted 2022-05-04 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Phase 2; SRF388; IL-27; safety; efficacy; immunotherapy; cancer; immuno-oncology; liver cancer; hepatocellular carcinoma; atezolizumab; Tecentriq; bevacizumab; Avastin
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms; Liver Neoplasms | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lead-In (Experimental): A minimum of 6 patients and up to 30 patients will be enrolled in an open-label Lead-In to assess the preliminary safety and tolerability of SRF388 with atezolizumab plus bevacizumab.
  Interventions: Drug: SRF388; Drug: Atezolizumab; Drug: Bevacizumab
- Arm A: SRF388 in Combination with atezolizumab plus bevacizumab (Experimental): Patients randomized to Arm A will receive SRF388 with atezolizumab plus bevacizumab.
  Interventions: Drug: SRF388; Drug: Atezolizumab; Drug: Bevacizumab
- Arm B: Placebo in combination with atezolizumab plus bevacizumab (Experimental): Patients randomized to Arm B will receive placebo with atezolizumab plus bevacizumab.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Placebo

INTERVENTIONS:
Drug: SRF388 — SRF388 will be administered by intravenous injection (IV)
  Arms: Arm A: SRF388 in Combination with atezolizumab plus bevacizumab; Lead-In
Drug: Atezolizumab — Azezolizumab will be administered by IV
  Other Names: Tecentriq
Drug: Bevacizumab — Bevacizumab will be administered by IV
  Other Names: Avastin
Drug: Placebo — Placebo will be administered by IV
  Arms: Arm B: Placebo in combination with atezolizumab plus bevacizumab

SUMMARY:
This is a Phase 2 trial composed of an open label Lead-In followed by a Randomized Phase designed to evaluate the efficacy and safety of SRF388 in combination with atezolizumab plus bevacizumab compared to placebo (inactive substance) in combination with atezolizumab plus bevacizumab in patients with first-line advanced or metastatic HCC.

DETAILED DESCRIPTION:
This is a Phase 2 trial designed to evaluate the efficacy and safety of SRF388 in combination with atezolizumab plus bevacizumab (Arm A) compared to placebo in combination with atezolizumab plus bevacizumab (Arm B) in patients with first-line advanced or metastatic HCC.

After a Lead-In Phase of up to 30 patients who will receive open-label SRF388 + atezolizumab + bevacizumab, the blinded Randomized Phase will randomize approximately 104 patients with a 1:1 allocation to Arm A or Arm B and stratified by geographic region (Asia excluding Japan vs. rest of world) and Barcelona Clinic Liver Cancer (BCLC) stage (B or C).

ELIGIBILITY:
Abbreviated Inclusion Criteria:

* ≥ 18 years of age on day of signing informed consent
* Unresectable locally advanced or metastatic HCC
* No prior systemic treatment for unresectable locally advanced or metastatic HCC
* BCLC Stage B or Stage C disease
* Child-Pugh Class A disease
* ≥ 1 measurable lesion per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Laboratory values indicative of adequate organ function as defined in the protocol
* Women of childbearing potential must have a negative pregnancy test within 1 week prior to first dose of study drug
* Women of childbearing potential or men with a heterosexual partner of childbearing potential or pregnant must agree to refrain from sexual intercourse or be willing to use effective methods of contraception as defined in the protocol while receiving study drug and for 6 months after the last dose of any study drug

Abbreviated Exclusion Criteria:

* Currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Previously received an anti-interleukin (IL)-27 antibody (Ab) or anti-IL-27-targeted therapy.
* Received prior systemic therapy for unresectable or metastatic disease. (Note: Prior systemic therapies administered for neoadjuvant, adjuvant, or curative intent (localized disease) are permitted if they were given > 1 year prior to the development of recurrent or metastatic disease)
* Known fibrolamellar HCC histology, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Moderate or severe ascites
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* History of or current hepatic encephalopathy
* Unable to undergo disease evaluation with a triphasic CT or MRI because of contrast allergy or other contraindication
* Untreated or incompletely treated varices with bleeding or high risk for bleeding.
* Symptomatic or untreated brain metastases or leptomeningeal carcinomatosis.
* Active or history of autoimmune disease or immune deficiency with some exceptions such as controlled thyroid disease, Type 1 diabetes, eczema and other minor skin disorders.
* Medical conditions requiring chronic steroid therapy (ie, > 10 mg/day of prednisone or its equivalent) or anticipates the need for systemic immunosuppressive medications during treatment with study drug
* Known active infection with HIV
* Known infection with hepatitis B virus (HBV) or hepatitis C virus (HCV), except for controlled active HBV or fully treated HCV infection as defined by the protocol
* Inadequately controlled arterial hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Nature, frequency, and severity of adverse events (AEs) per NCI CTCAE version 5.0 or higher | Up to 2 years
  Summaries of AEs will be based on TEAEs. A TEAE is an AE that emerges or worsens in the period from the first dose of study drug to 30 days after the last dose of study drug (Lead-In Phase).
Progression Free Survival (PFS) according to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1) | Up to 2 years
  PFS according to RECIST v1.1 will be evaluated in patients receiving SRF388 in combination with atezolizumab plus bevacizumab compared to placebo in combination with atezolizumab plus bevacizumab (Randomized Phase).

SECONDARY OUTCOMES:
Progression Free Survival (PFS) according to RECIST v1.1 | Up to 2 years
  Progression Free Survival (PFS) according to RECIST v1.1 (Lead-In Phase).
PFS according to HCC modified RECIST (mRECIST) | Up to 2 years
  PFS according to HCC mRECIST.
Objective Response Rate (ORR) according to RECIST v1.1 | Up to 2 years
  ORR according to RECIST v1.1.
ORR according to HCC mRECIST | Up to 2 years
  ORR according to HCC mRECIST.
Duration of Response (DoR) according to RECIST 1.1 | Up to 2 years
  DoR will be determined according to RECIST v1.1.
Duration of Response (DoR) according to HCC mRECIST | Up to 2 years
  DoR will be determined according to HCC mRECIST.
Disease Control Rate (DCR) | Up to 2 years
  DCR will measure the proportion of patients who experience best overall response of complete response (CR), partial response (PR), or stable disease (SD).
Time to Progression (TTP) according to RECIST v1.1 | Up to 2 years
  TTP according to RECIST v1.1.
TTP according to mRECIST | Up to 2 years
  TTP according to HCC mRECIST.
Overall Survival (OS) | Up to 2 years
  OS, defined as time from study drug initiation (Lead-In) or randomization to death from any cause.
Time to Response according to RECIST v1.1 | Up to 2 years
  Time to response will be evaluated according to RECIST v1.1
Time to Response according to HCC mRECIST | Up to 2 years
  Time to response will be evaluated according to HCC mRECIST
Nature, frequency, and severity of adverse events (AEs) per NCI CTCAE version 5.0 or higher | Up to 2 years
  Summaries of AEs will be based on TEAEs. A TEAE is an AE that emerges or worsens in the period from the first dose of study drug to 30 days after the last dose of study drug (Randomized Phase).
Incidence of SRF388 Antidrug Antibodies (ADAs) | Up to 2 years
  Percentage of patients who develop ADAs to SRF388.
Incidence of atezolizumab ADAs | Up to 2 years
  Percentage of patients who develop ADAs to atezolizumab.
Maximum observed serum concentration (Cmax) of SRF388 | Up to 2 years
  Serum samples will be collected and analyzed to assess the Cmax of SRF388.
Time of maximum observed serum concentration (tmax) of SRF388 | Up to 2 years
  Serum samples will be collected and analyzed to assess the (tmax) of SRF388.
Area under the serum concentration-time curve from time zero to the last quantifiable time point (AUC0-last) | Up to 2 years
  Serum samples will be collected and analyzed to assess AUC0-last of SRF388.
Terminal elimination half-life (t1/2) | Up to 2 years
  Serum samples will be collected and analyzed to assess the t1/2 of SRF388.
Serum concentrations of atezolizumab | Up to 2 years
  Serum samples of atezolizumab will be collected to assess maintenance concentrations of atezolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Koho Iizuka, MD, Study Chair — Coherus Oncology, Inc.
Locations (37):
- United States (15):
  - University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - City of Hope, Duarte, California
  - University of Southern California - Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Louisville VA Medical Center - Robley Rex VA Medical Center, Louisville, Kentucky
  - Veterans Affairs Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan Health System (UMHS), Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Veterans Affairs New York Harbor Healthcare System - Manhattan VA Medical Center, New York, New York
  - NYU Langone Medical Center - Laura and Isaac Perlmutter Cancer Center (NYU Cancer Institute (NYUCI)), New York, New York
  - University of Oklahoma Health Sciences Center - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Sarah Cannon Research Institute - Tennessee Oncology, Chattanooga, Tennessee
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
- Australia (4):
  - The Alfred Hospital, Melbourne
  - Royal Melbourne Hospital, Melbourne
  - St George Hospital -Kogarah, NSW
  - Gold Coast Private Hospital, Southport
- South Korea (12):
  - The Catholic University of Korea - St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Daegu Catholic University Medical Center (DCUMC), Daegu
  - Chonnam National University (CNU) - Chonnam National University Hwasun Hospital (CNUHH), Gwangju
  - Ajou University Hospital, Gyeonggi-do
  - CHA University - Bundang CHA General Hospital (CHA Bundang Medical Center), Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam
  - Severance Hospital, Seoul
  - Gangnam Severance Hospital - Cancer Hospital, Seoul
  - Korea University Medical Center - Korea University Anam Hospital, Seoul
  - University of Ulsan College of Medicine - Asan Medical Center (AMC), Seoul
  - Seoul National University Hospital (SNUH) - SMG-SNU Boramae Medical Center, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Taiwan (6):
  - Buddhist Tzu Chi General Hospital - Hualien Tzu Chi Medical Center, Hualien City
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Cancer Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No